CLINICAL TRIAL: NCT03070093
Title: A Multicenter, Open-label Treatment Protocol of Gilteritinib (ASP2215) in Patients With FMS-like Tyrosine Kinase 3 (FLT3) Mutated Relapsed or Refractory Acute Myeloid Leukemia (AML) or FLT3-Mutated AML in Complete Remission (CR) With Minimal Residual Disease (MRD)
Brief Title: Expanded Access Study of Gilteritinib (ASP2215) in Patients With FMS-like Tyrosine Kinase 3 (FLT3) Mutated Relapsed or Refractory Acute Myeloid Leukemia (AML) or FLT3-Mutated AML in Complete Remission (CR) With Minimal Residual Disease (MRD)
Status: Approved for marketing | Type: Expanded Access
Sponsor: Astellas Pharma Global Development, Inc. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Other Study IDs: 2215-CL-9100
Record Dates: First submitted 2017-02-28; First posted 2017-03-03 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: Acute Myeloid Leukemia (AML); FMS-like Tyrosine Kinase-3 (FLT3) Mutations
Keywords: Acute myeloid leukemia (AML); FMS-like Tyrosine kinase-3 (FLT3) mutations; gilteritinib; Expanded access; ASP2215
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — gilteritinib

STUDY DESIGN:
Expanded Access Types: Treatment

INTERVENTIONS:
Drug: gilteritinib — oral
  Other Names: ASP2215

SUMMARY:
The purpose of this study is to provide expanded access to ASP2215 for subjects with FLT3-mutated relapsed or refractory AML or FLT3-mutated AML in composite complete remission (CRc) (complete remission [CR], complete remission with incomplete hematologic recovery [CRi], complete remission with incomplete platelet recovery [CRp]) with MRD without access to comparable or alternative therapy.

DETAILED DESCRIPTION:
The United States Food and Drug Administration (FDA), the Japanese Ministry of Health, Labour and Welfare (MHLW) and Health Canada have approved ASP2215/Gilteritinib (XOSPATA®) for the treatment of adult patients who have relapsed or refractory acute myeloid leukemia (AML) with a FLT3 mutation.

This treatment protocol is being conducted while phase 3 ASP2215 studies are ongoing in FLT3-mutated AML subjects.

Subjects will complete visits on cycle 1 - days 1, 4, 8, 15; cycle 2 - days 1, 15; cycles 3 to 6 - day 1; and day 1 of every 2 cycles thereafter (i.e., cycle 8 day 1, cycle 10 day 1, etc.) until discontinued from the study.

Subjects will be provided with study medication until the investigator determines the subject is no longer receiving clinical benefit.

An end of treatment visit will be performed within 7 days after last dose of investigational product (ASP2215), or prior to initiation of another anticancer therapy, whichever occurs earlier, followed by a 30-day follow-up. [Specific to investigational sites in Japan: Study population does not include subjects with FLT3-mutated AML in CRc (CR, CRi, CRp) with MRD. Hence, efficacy (MRD response rate and duration of response) data will not be collected for subjects enrolled in Japan.]

ELIGIBILITY:
Inclusion Criteria:

* Subject is considered an adult according to local regulation at the time of signing informed consent.
* Subject has a diagnosis of primary AML or AML secondary to myelodysplastic syndrome (MDS) or therapy-related AML according to World Health Organization (WHO) classification.
* Subject has presence of the FLT3-mutated relapsed or refractory AML or FLT3-mutated AML in CRc (CR, CRi, CRp) with MRD in bone marrow or peripheral blood. [Specific to investigational sites in Japan: FLT3-mutated AML in CRc (CR, CRi, CRp) with MRD subjects will not be included.]
* Subject has refractory or relapsed AML (with or without hematopoietic stem cell transplant [HSCT]) or AML in CRc (CR, CRi, CRp) with MRD by flow cytometry or genetic testing for the FLT3 mutation after induction/consolidation regimen or HSCT. [Specific to investigational sites in Japan: FLT3-mutated AML in CRc (CR, CRi, CRp) with MRD subjects will not be included.]
* Subject must wait for at least 5 half-lives after stopping therapy with any investigational agent and before starting ASP2215.
* Subject must meet the following criteria as indicated on clinical laboratory tests:

  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3x institutional upper limit of normal (ULN)
  * Serum total bilirubin ≤ 2.5 mg/dL, except for subjects with Gilbert's syndrome
  * Serum potassium and serum magnesium ≥ institutional lower limit of normal (LLN).
* Subject is able to tolerate oral administration of study drug.
* Subject who has developed overall grades II-IV acute graft-versus-host disease (GVHD) must satisfy the following criteria:

  * No requirement of > 0.5 mg/kg of prednisone (or equivalent) daily dose within 1 week of enrollment
  * No escalation of immunosuppression in terms of increase of corticosteroids or addition of new agent/modality in prior 2 weeks (note that increasing calcineurin inhibitors or sirolimus to achieve therapeutic trough levels is allowed)
* Female subject must either:

  * Be of nonchildbearing potential:
  * Postmenopausal (defined as at least 1 year without any menses) prior to screening, or
  * Documented surgically sterile (e.g., hysterectomy, bilateral salpingectomy, bilateral oophorectomy) at least 1 month prior to screening.
  * Or, if of childbearing potential,
  * Agree not to try to become pregnant during the study and for at least 180 days after the final study drug administration
  * And have a negative urine pregnancy test at screening
  * And, if heterosexually active, agree to use consistently 2 forms of effective contraception per locally accepted standards (1 of which must be a barrier method) starting at screening and throughout the study period and for at least 180 days after the final study drug administration.
* Female subject must agree not to breastfeed or donate ova starting at screening and throughout the study period, and for at least 180 days after the final study drug administration.
* Male subject (even if surgically sterilized) and partners who are women of childbearing potential must agree to practice 2 forms of effective contraception per locally accepted standards

  (1 of which must be a barrier method), starting at screening and throughout the study period and for 120 days after the final study drug administration.
* Male subject must not donate sperm starting at screening and throughout the study period and for 120 days after the final study drug administration.
* Subject agrees not to participate in another interventional study for AML while on treatment.
* Subject who has a diagnosis of HIV may be enrolled as long as the disease is under control on antiretroviral therapy. Precautions should be taken to modify highly active antiretroviral therapy (HAART) regimen to minimize drug interactions.
* There is no comparable or satisfactory alternative therapy to treat the subject's AML.

Exclusion Criteria:

* Subject is eligible to participate in an ongoing clinical study of ASP2215; or has previously participated in a randomized clinical study of ASP2215 with a primary endpoint of overall survival that is not closed for efficacy.
* Subject with QTcF > 450 ms at screening based on local reading.
* Subject with a known history of Long QT Syndrome at screening.
* Subject was diagnosed with acute promyelocytic leukemia (APL).
* Subject has BCR-ABL-positive leukemia (chronic myelogenous leukemia in blast crisis).
* Subject has clinically significant coagulation abnormality unless secondary to AML.
* Subject has active hepatitis B or C or an active hepatic disorder.
* Subject has uncontrolled angina, severe uncontrolled ventricular arrhythmias, electrocardiographic evidence of acute ischemia, or New York Heart Association (NYHA) Class IV heart failure.
* Subject requires treatment with concomitant drugs that are strong inducers of CYP3A.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has hypersensitivity to any of the study drug components.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development, Inc.
Locations (39):
- United States (32):
  - UCLA, Los Angeles, California
  - Rocky Mountain Cancer Center-M, Aurora, Colorado
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Northside Hospital, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northwestern University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation at Franciscan Health Indianapolis, Indianapolis, Indiana
  - Norton Cancer Institute, Louisville, Kentucky
  - Tulane University, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - Johns Hopkins Hospital, Baltimore, Maryland
  - The Sidney Kimmel Comprehensive Cancer Center -Johns Hopkins University, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - West Michigan Regional Cancer Center, Kalamazoo, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Roswell Park Cancer Institute, Buffalo, New York
  - Memorial Sloan Kettering, New York, New York
  - Weill Cornell Medical College, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest Baptist Hospital, Winston-Salem, North Carolina
  - Ohio State University, Columbus, Ohio
  - Providence Portland Medical Center, Portland, Oregon
  - Penn State Hershey Medical Center, Hershey, Pennsylvania
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - UPCI, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah
  - WVU Medicine Cancer, Morgantown, West Virginia
- Canada (4):
  - Site CA15002, Halifax, Nova Scotia
  - Site CA15003, Toronto, Ontario
  - Site CA15001, Montreal, Quebec
  - Site CA15005, Vancouver
- Japan (3):
  - Site JP81001, Nagoya, Aichi-ken
  - Site JP81002, Shinagawa-ku, Tokyo
  - Site JP81003, Fukuoka